CLINICAL TRIAL: NCT05687656
Title: A Prospective, Multi-center Observational Study to Investigate the Safety and Effectiveness of Sterilized, Porcine Placental Tissue in the Treatment of Chronic Diabetic Foot Ulcers
Brief Title: Sterilised, Porcine Placental Tissue in the Treatment of Chronic Diabetic Foot Ulcers
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: ConvaTec Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: TLS-IM-001
Record Dates: First submitted 2022-12-02; First posted 2023-01-18 (Actual); Last update posted 2025-05-31 (Actual); Status verified 2025-05

CONDITIONS: Diabetic Foot Ulcer
MeSH Terms: conditions — Diabetic Foot

STUDY DESIGN:
Intervention Model Description: Eligible subjects will be treated with a weekly application for 12 weeks of sterilized, porcine placental ECM followed by standard of care wound therapy and offloading
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (1):
- InnovaMatrix AC porcine placental ECM therapy (Experimental): Eligible subjects will be treated with a weekly application of sterilized, porcine placental ECM followed by standard of care wound therapy and offloading
  Interventions: Device: InnovaMatrix AC porcine placental ECM therapy

INTERVENTIONS:
Device: InnovaMatrix AC porcine placental ECM therapy — All eligible subjects will be treated with a weekly application of sterilized, porcine placental ECM followed by standard of care moist wound therapy and offloading

SUMMARY:
A Prospective, Non-Randomized, Multi-Center Observational Study

To determine the safety and effectiveness of InnovaMatrix AC porcine placental ECM therapy for the treatment of chronic, non-healing diabetic foot ulcers (DFUs)

Eligible subjects will be treated with a weekly application of sterilized, porcine placental ECM followed by standard of care wound therapy and offloading

DETAILED DESCRIPTION:
This is a prospective, multi-center observational study . The trial will include 30 completed subjects at three (3) experienced clinical centers in the United States. The estimated enrollment period is 13 weeks. After completing a screening , the subjects will be enrolled and receive treatment followed for at least 12 weeks.

It is expected that the majority of the subjects will be recruited from patients being seen in the Investigators' practices. No minors will be included in the study and it is anticipated that there will be a roughly equal representation of male and female subjects. Further, no subjects will be excluded because of race or ethnicity and all efforts will be made to adequately represent the study population in the area in which they are chosen.

All subjects will be used for the analysis of efficacy and safety data.

ELIGIBILITY:
Inclusion Criteria

1. Male or female patients over 18 years of age who have given written informed consent in accordance with the ICH Good Clinical Practice (GCP) guideline. Female subjects must be either of non-childbearing potential or if of child bearing potential must satisfy the defined contraceptive criteria Exclusion criteria h.
2. Patients who are willing and able to attend all follow up visits
3. Subject has a known history of Type 1 or Type 2 diabetes with a HbA1c ≤12% . Has a diabetic foot ulcer classified by the Wagner classification 1 or 2 and at least 0.75cm2 and less than 5.0 cm2 in surface area as determined by photographic planimetry at the time of enrollment.
4. Index ulcer characteristics:

   1. Ulcer present for ≥ 30 days prior to (Day 0)
   2. Index ulcer is located below the ankle: at least 50% of the ulcer surface area is below the malleolus.
5. Subject has Body Mass Index (BMI) ≤ 45 at enrollment.
6. Subject has adequate circulation to the affected extremity, as demonstrated by at least one of the following within the past 30 days:

   * Dorsum transcutaneous oxygen test (TcPO2) with results ≥ 30 mmHg, Or
   * ABIs with results of ≥ 0.7 and ≤ 1.2, Or
   * Doppler arterial waveforms, which are triphasic or biphasic at the ankle of the affected foot. For ABPI >1.2 TBI (Toe Brachial Index) > 0.5.
   * Patient able to ambulate at home or in the clinic with or without mobility aids

8. The subject is willing to accept treatment with a porcine based product 9. The subject is medically stable, in the opinion of the investigator

Exclusion Criteria:

1. Index Ulcer Assessment:

   1. Penetrates down to muscle, tendon, or bone
   2. Presence of another diabetic foot ulcer within 2 cm of the index ulcer
   3. Index ulcer determined to be due to Active Charcot deformity or previous surgical correction for Charcot deformity.
   4. Wounds which occur in relation to major structural abnormalities of the foot, which would include amputations related to osteomyelitis or Charcot deformity
   5. Exhibits overt clinical signs and symptoms of infection with cellulitis surrounding the wound margin.
   6. Known or suspected local skin malignancy to the index diabetic ulcer
   7. Wound duration > one year without intermittent closure
2. Prior therapies - Subjects receiving treatment with any of the following will not be eligible for enrollment:

   1. In the last 7 days - Negative pressure wound therapy (wound vac or SNaP®) of the index ulcer
   2. In the last 7 days - Hyperbaric oxygen (HBO) therapy
   3. In the last 10 days - Chemical debridement, hypochlorous acid or Dakin's solution, medical honey therapy
   4. In the last 30 days - Treatment with cytotoxic chemotherapy, application of topical steroids to the ulcer surface, or use of ≥ 14 days of immune-suppressants (including systemic corticosteroids); or, subject is anticipated to require such medications during the course of the study
   5. In the last 30 days - study ulcer treatment with any advanced therapy, including, biomedical or topical growth factors, tissue engineered materials (e.g. Apligraf or Dermagraft), sterilized placental allografts (EpiFix, NovaFix, etc.), or other scaffold materials (e.g. OASIS® Wound Matrix, MatriStem Wound Matrix )
   6. In the last 30 days - Subject has been on any investigational drug(s) or therapeutic device(s)
   7. In the last 8 weeks - Amputation or revascularization (surgical or stenting) to the affected leg
3. Subject criteria that will make subject ineligible for enrollment:

   1. Known hypersensitivity to porcine based products
   2. Known osteomyelitis or active cellulitis requiring antimicrobial therapy at wound site
   3. End stage renal disease requiring dialysis.
   4. Immune system disorders including Systemic Lupus Erythematosus (SLE), Acquired Immunodeficiency Syndrome (AIDS) or HIV
   5. Presence of any condition (including current drug or alcohol abuse, medical or psychiatric condition) that is likely to impair understanding of or compliance with the study protocol in the judgment of the Investigator
   6. Pregnancy at enrollment or within last 6 months, women who are breastfeeding, or women of childbearing potential who are planning to become pregnant during the time of the study OR are unwilling/unable to use acceptable methods of contraception (birth control pills, barriers, or abstinence)
   7. Subjects currently enrolled in this study. Concurrent enrollment in the study is prohibited
   8. Subjects currently receiving radiation therapy or chemotherapy
   9. Any pathology that would limit the blood supply and compromise healing or non-revascularizable surgical sites

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2022-10-06 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Wound Healing area using digital image | 12 weeks
  The primary endpoint for the study is assessment of ulcer area at Weeks 6 and 12 using the MolecuLight Imaging Device

SECONDARY OUTCOMES:
Wound Closure | 12 weeks
  Time to complete wound closure as defined by FDA
Percentage area reduction | 12 weeks
  • Rate of wound closure as assessed by wound area measurements determined by weekly percent area reduction
Adverse events | 12 weeks
  Adverse events as reported at weekly treatment visits

OTHER OUTCOMES:
Bacterial burden assessment | 12 weeks
  Reduction in bacterial burden as assessed by fluorescence imaging using the moleculight imaging device at weeks 4, 8 and 12.
Presence of protease levels | 12 weeks
  Reduction in host proteases at weeks 4,8, and 12.

CONTACTS AND LOCATIONS:
Overall Officials: Thomas E Serena, MD, Principal Investigator — SerenaGroup, Inc.
Locations (5):
- United States (5):
  - Three Rivers Hyperbaric and Wound Center, North Port, Florida
  - Serena Group Buffalo Research Center, Buffalo, New York
  - SerenaGroup Monroeville, Monroeville, Pennsylvania
  - SerenaGroup Austin Research Center, Austin, Texas
  - Atrium Medical Center, Stafford, Texas